CLINICAL TRIAL: NCT01352104
Title: Effectiveness of Guiding Teachers in Individualized Behavioral Intervention Strategies With Preschool Children Indicated for Externalizing Problem Behavior
Brief Title: Effectiveness of the Teacher Module of the Prevention Program for Externalizing Problem Behaviour in Preschoolers
Acronym: PEP-TE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Research Foundation (Other)
Responsible Party: Manfred Döpfner, Clinic of Child and Adolescent Psychiatrie and Psychotherapy, University of Cologne, Germany
Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DO 620/2-4
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-04

CONDITIONS: Behavior Problem of Childhood and Adolescence
Keywords: Externalizing Problem Behaviour in Preschoolers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- waiting-intervention-course (Experimental)
  Interventions: Behavioral: PEP-TE

INTERVENTIONS:
Behavioral: PEP-TE — PEP-TE for kindergarten teachers of children with externalizing behaviour problems aged 3 to 6 years leads to use classical strategies of changing behaviour (defining rules, appropriate commands, positive and negative consequences) based on the "coercive interaction process" (cf. Patterson, 1982) as explanatory model for target situations. In 10 units (90-120 minutes) four to six teachers in one group develop individually tailored solutions to specified externalizing behavior problems of the target child. General strategies of improving positive interactions as well as resources and strategies for reducing stress and gaining new energy are discussed. Summary and reflection of the teacher' experiences and ideas of changes in routines prevents relapses.

SUMMARY:
Investigating effectiveness of the cognitive-behavioral based teacher training under routine care conditions by comparison of a baseline-interval with no special intervention to a following interval of PEP for the kindergarten teachers only each focussing on one child (3-6 years old) that the teacher herself indicated as "needing special attention for externalising behaviour". Effects on child symptoms and teachers behavior and burden within intervention-period are expected to be stronger than those during waiting-period.

DETAILED DESCRIPTION:
Findings of the PEP-efficacy-study based on a randomised controlled sampling ((ISRCTN CCT-NAPN-18918) using combined training-modules for parents and teachers showed positive effects on children's behaviour in the intervention-group. These effects in teacher's view were stronger than in the control-group but could not be proved to be statistically significant. Moreover after this first step of evaluation there remain unanswered questions concerning the stability of effects after transferring the program in routine care. Therefore the study is continued by an effectiveness-study.

ELIGIBILITY:
Inclusion Criteria:

* teacher's interest in participating in a specific further training
* Identification of a target child (externalizing problem behavior)by teacher
* possibility of participation in at least 4 assessments (pre1, pre2, post,1stFU)

Exclusion Criteria:

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in children's externalizing behavior | pre1, pre2, post, 3-, 6-, 9- & 12 month FU
  Externalizing Behavior Scale of the Caregiver/Teacher-Report Form (C-TRF/ 1 1/2-, Achenbach, T.M. & Rescorla L.A.,2001) rated by participating teacher

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Döpfner, PhD, Principal Investigator — University of Cologne
Locations (1):
- Clinic for Child and Adolescent Psychiatry and Psychotherapy, University of Cologne, Cologne, North Rhine-Westphalia, Germany